CLINICAL TRIAL: NCT01002729
Title: Oseltamivir Pharmacokinetics in Morbid Obesity
Acronym: OPTIMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Canadian Center for Vaccinology (Other); Nova Scotia Health Authority (Other); Dalhousie University (Other); Hoffmann-La Roche (Industry)
Responsible Party: McNeil, Shelly, IWK Health Sciences Center / Capital Distict Health Authority
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC91
Record Dates: First submitted 2009-10-25; First posted 2009-10-27 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Morbid Obesity
Keywords: Oseltamivir Pharmacokinetics Obesity; Oseltamivir Pharmacokinetics in Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patients with a BMI < 30 given Oseltamivir — Patients with a BMI < 30 given Oseltamivir
Other: Patients with a BMI > 40 given Oseltamivir — Patients with a BMI > 40 given Oseltamivir

SUMMARY:
This trial asks the question: do people of much greater than average body weight need more of a drug called oseltamivir than current recommendations suggest. Oseltamivir is a drug given to people who have influenza, and currently is also being used to fight the new H1N1 influenza. Some people of larger than average body weight require larger amounts of drugs to see the same effects as others of an average body weight. No studies have ever been conducted looking at the possibility of oseltamivir being one of those drugs. Our Study's hypothesis states that those of an above average body weight will have different amounts of drug in their blood than those of people of normal body weight if they are given the normal amount prescribed for influenza. Our study will give oseltamivir to twenty people for 7 days. Half of the people will be of normal body weight and the others will be of a much higher than normal body weight. Using blood samples the investigators will determine if the amounts of oseltamivir are significantly lower in the blood of patients in the above normal body weight group.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 55 years
* Written informed consent
* Subjects without medical history, physical finding or laboratory finding, which, in the opinion of the investigator, could pose a safety concern or interfere with the protocol.

Exclusion Criteria:

* Allergy to oseltamivir
* Blood donation within 3 months before oseltamivir administration
* Medications that may interfere with the disposition of oseltamivir (e.g. probenecid)
* Anemia
* Estimated Creatinine clearance < 60 ml/min (As calculated by the modified Cockcroft Gault equation below) Creatinine Clearance= (140-Age) x 1.2 x Adjusted Body weight (x 0.85 if female) Serum Creatinine (umol/L)

Adjusted body weight = Ideal body weight + [0.4 (Actual Bodyweight-Ideal Body Weight)]

* Gastrectomy
* Enterectomy (or any other surgical procedure that would interfere with absorption)
* Clinically significant haematological (RBC count, WBC count, WBC differential count, platelets count and haemoglobin level) or biochemical (ALT, AST, creatinine and urea) abnormalities as per the judgement of the investigator
* Clinically significant cardiac conduction abnormality noted on baseline electrocardiogram.
* Influenza like illness (fever and/or cough plus one of the following sore throat, fatigue, myalgia, headache) within 7 days of enrolment
* Pregnancy
* Inability to consume study meals provided due to special dietary requirements such as food allergies.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Serum Drug Concentration | 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Lucas M Thorne-Humphrey, BSC Pharm, Study Chair — Dalhousie Unviersity, Captial District Health Authority
Locations (1):
- Human Vaccine Challenge Unit, IWK Health Center, Halifax, Nova Scotia, Canada

REFERENCES:
- [Result] Thorne-Humphrey LM, Goralski KB, Slayter KL, Hatchette TF, Johnston BL, McNeil SA; 2009 OPTIMO Study Group. Oseltamivir pharmacokinetics in morbid obesity (OPTIMO trial). J Antimicrob Chemother. 2011 Sep;66(9):2083-91. doi: 10.1093/jac/dkr257. Epub 2011 Jun 23. PMID 21700623